CLINICAL TRIAL: NCT04618510
Title: Efficacy of SEED's Novel Anti-myopia Contact Lens (Daily Disposable) in Controlling Myopia Progression
Brief Title: SEED-LVPEI Myopia Study
Acronym: SLIMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: L.V. Prasad Eye Institute (Other)
Collaborators: SEED Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Dr. Pavan Verkicharla, Scientist-Myopia Research Lab, L.V. Prasad Eye Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEC-BHR-P-09-20-511
Record Dates: First submitted 2020-10-27; First posted 2020-11-06 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Myopia
Keywords: Myopia; Contact Lens; Peripheral Defocus; Multi-focal; India; Extended Depth of Focus
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Masked Randomized Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEED 1-dayPure EDOF soft contact lens (Experimental): The participant will be requested to wear the daily disposable lens 8-10 hours per day and replaced daily. All participants will be followed for 12 months (followup visit schedule; 3 months, 6 months, 12 months) post-contact lens wear.
  Interventions: Device: SEED 1-dayPure EDOF soft contact lens
- Single vision spectacle lens (Sham Comparator): The participant will be requested to wear the spectacle lens daily. All participants will be followed for 12 months (follow up visit schedule; 3 months, 6 months, 12 months) post spectacle lens wear.
  Interventions: Device: Single Vision Spectacles

INTERVENTIONS:
Device: SEED 1-dayPure EDOF soft contact lens — Centre-distance contact lens with peripheral add power working on extended depth of focus principle to control myopia
  Arms: SEED 1-dayPure EDOF soft contact lens
Device: Single Vision Spectacles — These are the type of glasses that correct vision for a single distance
  Arms: Single vision spectacle lens

SUMMARY:
This randomized clinical trial study aims to investigate the efficacy of novel SEED's EDOF based mid-lens design in controlling the myopia progression in

Indian children with these specific objectives:

1. To investigate the efficacy of SEED's 1-day pure extended depth of focus lenses controlling myopia progression in Indian children through a one-year randomized clinical study.
2. To investigate the role of SEED's 1-day pure extended depth of focus lenses in altering peripheral refraction of the eye to control myopia progression.
3. To determine if there is any specific cohort that shows better efficacy in myopia control with 1-day pure extended depth of focus lenses based on central and peripheral optics (degree of myopia and optical parameters).
4. To investigate the qualitative assessment of comfort and visual experience with the SEED's EDOF contact lenses through the questionnaire method.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical trial will be conducted in Myopia Research Lab, L V Prasad Eye Institute, Hyderabad and the study protocol will adhere to the tenets of the Declaration of Helsinki. Participants will be recruited through advertisements in local print media (newspaper), approaching schools, through clinical referrals. Children will be assigned to either the control group or intervention group randomly based on computer-generated random numbers operated by the investigator. All participants will undergo a cycloplegic refractive error assessment after the instillation of tropicamide 1% eye drops (or cyclopentolate 1% eye drops in case of varying refractive error between objective and subjective values). Axial length and cycloplegic refractive measurements will be taken with using Lenstar LS900 biometer and Shin- Nippon autorefractor respectively for scheduled follow up and will be compared with the baseline parameters.

ELIGIBILITY:
Inclusion Criteria:

* Myopia (SE) between -0.50D to -10.00D
* Astigmatism less than 0.75D
* Anisometropia less than 1.00D
* Age of the participant from 7 to 15 years
* Neophyte or existing soft contact lens wearer
* Best-corrected visual acuity (BCVA); ≤ 20/20
* Participants who are willing to wear the contact lens constantly

Exclusion Criteria:

* Participants who had any ocular or systemic conditions that could influence the refractive error
* Poor compliance of contact lenses from existing wearer
* Prior use of orthokeratology lenses/bifocal lenses/anti-myopia strategies
* Participants who had any medications that could influence the refractive error

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Central refractive error changes | Data will be collected at baseline, 3 months, 6 months and 12 months.
  1. Changes (1 year) in spherical equivalent refractive error (dioptre) in the intervention and control group from the baseline.
  2. Changes (1 year) in spherical equivalent refractive error (dioptre) among different degrees of myopia in the intervention and control group from the baseline.
Axial length changes | Data will be collected at baseline, 3 months, 6 months and 12 months.
  1. Changes (1 year) in axial length (millimetre) in the intervention and control group from the baseline.
  2. Changes (1 year) in axial length (millimetre) among different degrees of myopia in the intervention and control group from the baseline.
Peripheral refractive error changes | Data will be collected at baseline, 3 months, 6 months and 12 months.
  1. Changes (1 year) in peripheral spherical equivalent refractive error (dioptre) of the individuals in the intervention and control group from the baseline.
  2. Changes (1 year) in peripheral spherical equivalent refractive error (dioptre) among different degrees of myopia in the intervention and control group from the baseline.

SECONDARY OUTCOMES:
Qualitative assessment | Data will be collected at 3 months, 6 months and 12 months.
  Qualitative assessment of discomfort and visual experience of centre-distance multifocal contact lens will be measured on a scale of 0-4 (0=Never, 1=Rarely, 2=Sometimes, 3=Often, 4=Always).

CONTACTS AND LOCATIONS:
Overall Officials: Pavan K Verkicharla, PhD, Principal Investigator — L.V. Prasad Eye Institute
Locations (1):
- Pavan K. Verkicharla, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sankaridurg P, Holden B, Smith E 3rd, Naduvilath T, Chen X, de la Jara PL, Martinez A, Kwan J, Ho A, Frick K, Ge J. Decrease in rate of myopia progression with a contact lens designed to reduce relative peripheral hyperopia: one-year results. Invest Ophthalmol Vis Sci. 2011 Dec 9;52(13):9362-7. doi: 10.1167/iovs.11-7260. PMID 22039230
- [Background] Bakaraju RC, Ehrmann K, Ho A. Extended depth of focus contact lenses vs. two commercial multifocals: Part 1. Optical performance evaluation via computed through-focus retinal image quality metrics. J Optom. 2018 Jan-Mar;11(1):10-20. doi: 10.1016/j.optom.2017.04.003. Epub 2017 Jun 9. PMID 28606456
- [Background] Bakaraju RC, Tilia D, Sha J, Diec J, Chung J, Kho D, Delaney S, Munro A, Thomas V. Extended depth of focus contact lenses vs. two commercial multifocals: Part 2. Visual performance after 1 week of lens wear. J Optom. 2018 Jan-Mar;11(1):21-32. doi: 10.1016/j.optom.2017.04.001. Epub 2017 Jun 12. PMID 28619486
- [Background] Sankaridurg P, Bakaraju RC, Naduvilath T, Chen X, Weng R, Tilia D, Xu P, Li W, Conrad F, Smith EL 3rd, Ehrmann K. Myopia control with novel central and peripheral plus contact lenses and extended depth of focus contact lenses: 2 year results from a randomised clinical trial. Ophthalmic Physiol Opt. 2019 Jul;39(4):294-307. doi: 10.1111/opo.12621. Epub 2019 Jun 10. PMID 31180155